CLINICAL TRIAL: NCT02972840
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study of Bendamustine and Rituximab (BR) Alone Versus in Combination With Acalabrutinib (ACP-196) in Subjects With Previously Untreated Mantle Cell Lymphoma
Brief Title: A Study of BR Alone Versus in Combination With Acalabrutinib in Subjects With Previously Untreated MCL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACE-LY-308; 2015-005220-26 (EudraCT Number)
Record Dates: First submitted 2016-11-21; First posted 2016-11-25 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma, Mantle Cell
Keywords: Bruton tyrosine kinase inhibitor; Acalabrutinib; Mantle Cell Lymphoma; ACE-LY-308; Treatment naive; non-Hodgkins Lymphoma; Bendomustine; Rituximab
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — acalabrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acalabrutinib in combination with bendamustine and rituximab (Experimental): Acalabrutinib administered twice per day (BID) orally (PO) plus bendamustine on Days 1 and 2 and rituximab on Day 1; cycles are repeated every 28 days.
  Interventions: Drug: Acalabrutinib; Drug: Bendamustine; Drug: Rituximab
- Placebo in combination with bendamustine and rituximab (Placebo Comparator): Matching placebo administered BID PO plus bendamustine on Days 1 and 2 and rituximab on Day 1; cycles are repeated every 28 days.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Placebo

INTERVENTIONS:
Drug: Acalabrutinib — Administered orally (PO)
  Other Names: ACP-196; Calquence
  Arms: Acalabrutinib in combination with bendamustine and rituximab
Drug: Bendamustine — Administered intravenously (IV)
  Other Names: Treanda; Bendeka
Drug: Rituximab — Administered intravenously (IV)
  Other Names: Rituxan; Rituxan Hycela
Drug: Placebo — Placebo comparator
  Arms: Placebo in combination with bendamustine and rituximab

SUMMARY:
This study is evaluating the efficacy of acalabrutinib in combination with bendamustine and rituximab (BR) compared with placebo plus BR in subjects with previously untreated mantle cell lymphoma.

DETAILED DESCRIPTION:
To evaluate the efficacy of acalabrutinib in combination with bendamustine and rituximab (BR) compared with placebo plus BR based on Independent Review Committee (IRC) assessment of progression-free survival (PFS) per the Lugano Classification for Non-Hodgkin Lymphoma (NHL) in subjects with previously untreated mantle cell lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ≥ 65 years of age.
* Pathologically confirmed MCL, with documentation of a chromosome translocation t(11;14)(q13;q32) and/or overexpression of cyclin D1 in association with other relevant markers (eg, CD5, CD19, CD20, PAX5) .
* MCL requiring treatment and for which no prior systemic anticancer therapies have been received.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Agreement to use highly effective forms of contraception during the study and 6 months after the last dose of bendamustine, or 12 months after the last dose of rituximab, whichever is longest .

Exclusion Criteria:

* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of first dose of study drug, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 480 msec (calculated using Friderica's formula: QT/RR0.33) at screening. Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening are allowed to enroll on study.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
* Uncontrolled active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment), or intravenous anti infective treatment within 2 weeks before first dose of study drug.
* Concurrent participation in another therapeutic clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 635 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival per the Lugano Classification for NHL in Arm 1 compared to Arm 2 | Up to 6 years
  Defined as the time from the date of randomization until disease progression (assessed by the IRC per the Lugano Classification for NHL) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Investigator-assessed progression-free survival per the Lugano Classification for NHL in Arm 1 compared to Arm 2 | Up to 6 years
  Defined as the time from the date of randomization until disease progression (assessed by the investigator per the Lugano Classification for NHL) or death from any cause, whichever occurs first.
Investigator-assessed overall response rate per the Lugano Classification for NHL in Arm 1 compared to Arm 2 | Up to 6 years
  Defined as the proportion of subjects who achieve either partial response (PR) or complete response (CR) as best overall response according to the Lugano Classification for NHL as assessed by investigator.
IRC-assessed overall response rate per the Lugano Classification for NHL in Arm 1 compared to Arm 2 | Up to 6 years
  Defined as the proportion of subjects who achieve either PR or CR as best overall response according to the Lugano Classification for NHL as assessed by IRC.
Overall survival in Arm 1 compared to Arm 2 | Up to 6 years
  Defined as the time from randomization until the date of death from any cause.
IRC-assessed duration of response per the Lugano Classification for NHL in Arm 1 compared to Arm 2 | Up to 6 years
  Defined as the time from the first documentation of CR or PR to disease progression per the Lugano Classification for NHL or death from any cause, whichever occurs first.
IRC assessed time to response per the Lugano Classification for NHL in Arm 1 compared to Arm 2 | Up to 6 years
  Defined as the time from randomization to the first CR or PR per the Lugano Classification for NHL.

CONTACTS AND LOCATIONS:
Locations (190):
- United States (30):
  - Research Site, Tucson, Arizona
  - Research Site, Downey, California
  - Research Site, Santa Monica, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Tallahassee, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Westwood, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Hawthorne, New York
  - Research Site, Lake Success, New York
  - Research Site, Portland, Oregon
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Fort Belvoir, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
- Argentina (3):
  - Research Site, Buenos Aires
  - Research Site, Caba
  - Research Site, Córdoba
- Australia (13):
  - Research Site, Bedford Park
  - Research Site, Concord
  - Research Site, Frankston
  - Research Site, Gosford
  - Research Site, Heidelberg
  - Research Site, Herston
  - Research Site, Kogarah
  - Research Site, Murdoch
  - Research Site, Nedlands
  - Research Site, Newcastle
  - Research Site, Southport
  - Research Site, Sydney
  - Research Site, Woolloongabba
- Belgium (5):
  - Research Site, Antwerp
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Roeselare
  - Research Site, Sint-Niklaas
- Brazil (7):
  - Research Site, Bela Vista
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, So Paulo
- Canada (6):
  - Research Site, Vancouver, British Columbia
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Edmonton
  - Research Site, Greenfield Park
  - Research Site, Halifax
- China (23):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Gongshu District
  - Research Site, Haidian District
  - Research Site, Harbin
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Tianjian
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuhou District
  - Research Site, Xicheng District
  - Research Site, Xuhui District
  - Research Site, Xuzhou
  - Research Site, Zhengzhou
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Ostrava Poruba
  - Research Site, Pilsen
  - Research Site, Prague
- France (9):
  - Research Site, Argenteuil
  - Research Site, Bobigny
  - Research Site, Bordeaux
  - Research Site, Le Mans
  - Research Site, Limoges
  - Research Site, Pessac
  - Research Site, Périgueux
  - Research Site, Rennes
  - Research Site, Vienne
- Germany (7):
  - Research Site, Heidelberg
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nordrhein-Westfalen
  - Research Site, Ravensburg
  - Research Site, Rheinland-Pfalz
  - Research Site, Ulm
- Greece (4):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Pok Fu Lam
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Pécs
  - Research Site, Szeged
- Israel (4):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
- Italy (8):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Reggio Emilia
  - Research Site, Rozzano
  - Research Site, Turin
- Japan (11):
  - Research Site, Fukuoka
  - Research Site, Kobe
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shimane
  - Research Site, Tokyo
  - Research Site, Yokohama
- Mexico (4):
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Querétaro
- New Zealand (3):
  - Research Site, Dunedin
  - Research Site, Grafton
  - Research Site, Otahuhu
- Peru (3):
  - Research Site, Arequipa
  - Research Site, Bellavista
  - Research Site, Lima
- Poland (8):
  - Research Site, Chorzów
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Warsaw
  - Research Site, Woj. Podkarpackie
  - Research Site, Wroclaw
- Romania (4):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Iași
- Russia (4):
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Syktyvkar
  - Research Site, Tula
- South Korea (3):
  - Research Site, Busan
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (7):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Ukraine (6):
  - Research Site, Cherkasy
  - Research Site, Chernihiv
  - Research Site, Dnipropetrovsk
  - Research Site, Kiev
  - Research Site, Lviv
  - Research Site, Zhytomyr
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements athttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Wang M, Salek D, Belada D, Song Y, Jurczak W, Kahl BS, Paludo J, Chu MP, Kryachok I, Fogliatto L, Cheah CY, Morawska M, Sancho JM, Li Y, Patti C, Forsyth C, Zhang J, Lesley R, Ramadan S, Rule S, Dreyling M; ECHO investigators; ECHO Investigators. Acalabrutinib Plus Bendamustine-Rituximab in Untreated Mantle Cell Lymphoma. J Clin Oncol. 2025 Jul 10;43(20):2276-2284. doi: 10.1200/JCO-25-00690. Epub 2025 May 1. PMID 40311141